CLINICAL TRIAL: NCT00178542
Title: Changes in Thrombin Generation Potential and Thromboelastography During the Menstrual Cycle
Brief Title: Change in Thrombin Generation Potential and Thromboelastography During the Menstrual Cycle
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The ZLB Behring Foundation (Unknown)
Responsible Party: Principal Investigator, Deborah Brown, Associate Profess - Gulf States Hemophilia Center, The University of Texas Health Science Center, Houston
Other Study IDs: TG and TEG
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Von Willebrand Disease
Keywords: von Willebrand Disease; Healthy Women and Women with von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to describe characteristics and trends for thrombin generation (TG) and thromboelastography (TEG) at 4 time points during the menstrual cycle.

DETAILED DESCRIPTION:
We propose that TG and TEG will be more sensitive than traditional coagulation assays to detect physiologic variation in hemostasis, fibrinolysis, and platelet activation throughout the menstrual cycle. We expect that TG and TEG will better discriminate patients with vWD than traditional coagulation studies during the menstrual cycle. In this study we plan to measure TG and TEG in healthy women and women with von Willebrand's disorder during four phases of the menstrual cycle. We will compare specific measurements of endogenous thrombin generation potential from the TG and fibrinolysis and platelet activation from the TEG with standard measures of coagulation, fibrinolysis, and platelet activation markers during the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Females of reproductive age with regular menstrual cycles and a diagnosis of von Willebrand disease according to the International Society of Thrombosis and Hemostasis diagnostic criteria.

Exclusion Criteria:

* Females who are pregnant, or have a history of endocrinopathy or hormone imbalance
* History of hysterectomy or bilateral oophorectomy
* History of ovarian or uterine cancer
* Use of intrauterine device
* Use of antifibrinolytic therapy, hemostatic agents, or anti-platelet agents.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females with a diagnosis of von Willebrand Disease
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Endogenous Thrombin Potential | 4 weeks
  Comparison of 4 values collected during 4 phases of through the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Brown, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States